CLINICAL TRIAL: NCT06765694
Title: Efficacy of One or Two Botulinum Toxin Injections in the Treatment of Chronic Lateral Epicondylalgia: a Retrospective Study
Brief Title: Efficacy of One or Two Botulinum Toxin Injections in the Treatment of Chronic Lateral Epicondylalgia: a Retrospective Study (EPITOX)
Acronym: EPITOX
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0278 - EPITOX
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-09

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- epicondylitis with BTX injection: Subjects included were addressed to a unique physician who performed all the treatment procedure with a diagnostic of lateral epicondylitis to receive a BTX injection.
  Interventions: Drug: Botulinum toxin injection

INTERVENTIONS:
Drug: Botulinum toxin injection — first injection was done under ultrasound control in the extensor carpi radialis brevis (ECRB). The second one if necessary was subordinated to clinical examination and focused in one or more of the following: ECRB, extensor digitorum communis, supinator.

SUMMARY:
Despite being a self-limiting injury, lateral epicondylitis (LE) can be difficult to manage. In cases of refractory LE, conservative treatment fails and symptoms persist over 6 months. Previous studies have investigated the role of botulinum Toxin Type A (BoNT-A) injections in LE with controversial results. There is some evidence that repeating the BoNT-A injection could be beneficial for refractory cases.

The objective is to assess the success rate of one or two BoNT-A injections for refractory LE.

ELIGIBILITY:
Inclusion Criteria:

lateral epicondylitis at least one botulinum injection

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects with chronic lateral epicondylitis already treated by physiotherapy, shock wave therapy, steroid injections without relief of pain
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
pain improvement | from enrollment to 6 months
  A qualitative scale was used to define the result of the treatment procedure based on pain improvement.
  Poor : no improvement Temporary : significant but temporary pain reduction Partial : permanent but partial pain reduction Good : patient no longer requesting any treatment for LE due to pain relief

SECONDARY OUTCOMES:
adverse events | from enrollment to 6 months
  Any adverse event was notified

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No